CLINICAL TRIAL: NCT04077281
Title: Improving Medication Prescribing-Related Outcomes for Vulnerable Elderly in Transitions (IMPROVE-IT): a Pilot Randomized Trial
Brief Title: Improving Medication Prescribing-Related Outcomes for Vulnerable Elderly in Transitions
Acronym: IMPROVE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Anne Holbrook, Director, Division of Clinical Pharmacology & Toxicology Professor, Department of Medicine, McMaster University Medical Staff, Hamilton Health Sciences and St Joseph's Healthcare Hamilton, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: CIHR#419518
Record Dates: First submitted 2019-08-07; First posted 2019-09-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Patient Discharge; Drug-Related Side Effects and Adverse Reactions; Aged; Health Care Costs
Keywords: Polypharmacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Clinical Pharmacology specialist team approach starting in hospital and following up with the patient at home using telemedicine and detailed communication with them, their caregiver, family physician, community pharmacist and other specialists.
  Interventions: Other: Medication Coordinated care
- Control Arm (Usual care) (No Intervention): Patients will receive a best possible medication history (BPMH) as do the intervention patients, then usual care by their primary team.

INTERVENTIONS:
Other: Medication Coordinated care — * Clinical Pharmacology & Toxicology consult
  * CPT team completes detailed circle of care communication
  * Telemedicine followup by CPT team (approximately 48 hrs post-discharge & 1 week to1 month post-discharge)
  Arms: Intervention Arm

SUMMARY:
Medication safety is a crucial health issue for every older Canadian since many of the medications causing serious harm are those which also have life-saving or important symptom-relieving benefits. Very few specialists can accurately advise seniors which medications provide more benefit than harm for them personally, and make changes safely as this requires a very large breadth and depth of knowledge about the patient, the conditions they have and their therapies. Now that telemedicine is compatible with smart phones, this extends the ability of scarce specialists to 'see' any patient in Canada in a way that is more convenient for the patient and may be less expensive than current care. This project will find out whether a unique Clinical Pharmacology specialist team in Hamilton, Ontario can improve medication safety (stop medications no longer needed, reduce doses where appropriate, change to safer medications) for a high risk group of older hospitalized Canadians taking many medications. The hospital where this pilot study will take place was the first to install the world's leading electronic health record and set it up to facilitate and support high quality research. Patients who volunteer will be assigned to their usual care, or to the intervention which is the Clinical Pharmacology specialist team approach starting in hospital and following up with the patient at home using telemedicine and detailed communication with them, their caregiver, family physician, community pharmacist and other specialists. The investigators will study whether the intervention is effective and cost-effective at reducing harmful medication burden, reducing the need to return to hospital, or improving the patient's ratings of their care coordination. The results will determine whether a subsequent large trial is worthwhile.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 65 years.
* Admitted to Medicine or Surgery services for more than 2 days.
* High cost users (defined as):
* Have at least one other hospitalization within the previous year.
* Taking 5 or more chronic medications including at least one TRIIM-Med.
* Provide informed consent.

Exclusion Criteria:

* Patients with "do not approach status".
* Patient or Caregiver not fluent in English.
* Patients who do not provide informed consent.
* Patients admitted for < 2 days.
* Patients < 65 years of age.
* Not a high cost user (as defined above).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcome: Recruitment rate for eligible patients. | Through the study completion, an average of 2 years
  The main trial will be considered feasible if we are able to recruit at least 50% of eligible patients in this pilot.
Clinical Outcome: The number of TRIIM-Meds successfully deprescribed. | 2 months post discharge
  The number of TRIIM-Meds successfully deprescribed (dose reduction or discontinued) at 2 months post-hospital discharge, aiming to be able to detect a mean difference of 0.5.

SECONDARY OUTCOMES:
Feasibility Outcomes of CPT consultation volume capacity and potential to apply the intervention entirely through telemedicine. | Through the study completion, an average of 2 years
  This will be measured based on the number of successfully enrolled patients, and the number of patients that will entirely undergo the intervention through telemedicine.
Feasibility Outcomes of patient retention rate. | Through the study completion, an average of 2 years
  This will be measured by looking at the number of patients enrolled, the number of patients that dropped out, and the number of patients that completed the study.
Feasibility Outcomes of likelihood of the intervention proving cost-effective. | Through the study completion, an average of 2 years
  This will be measured using Healthcare resource utilization questionnaire, which will determine whether the intervention reduced healthcare costs compared to the control group.
Patient-important outcomes: Participant ratings of coordination and continuity of transitions in care. | 2 months post discharge
  This outcome will be measured using the Coordination and Continuity of Care Questionnaire (CCCQ). Which is a questionnaire we adapted from the brief prepared questionnaire (B-PREPARED) and the three-question care transitions measure questionnaire (CTM-3).
Patient-important outcomes: Health related quality of life: EQ-5D-5L | 2 months post discharge
  This outcome will be measured using the EuroQol five-dimensional, five-level descriptive system (EQ-5D-5L) that asks patients to self-assess their own health quality related quality of life. Whereas a scoring metric is used to assess the overall health related quality of life based on the answers to the questions. The questionnaire scale considers 1 as the best possible health and 5 as the worst health possible.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Holbrook, Principal Investigator — St. Joseph's Healthcare Hamilton; Anne Holbrook, Principal Investigator — SJHH
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holbrook A, Perri D, Levine M, Mbuagbaw L, Jarmain S, Thabane L, Tarride JE, Dolovich L, Hyland S, Telford V, Silva J, Nieuwstraten C. Improving medication prescribing-related outcomes for vulnerable elderly in transitions on high-risk medications (IMPROVE-IT HRM): a pilot randomized trial protocol. Pilot Feasibility Stud. 2024 Apr 10;10(1):60. doi: 10.1186/s40814-024-01484-6. PMID 38600599